CLINICAL TRIAL: NCT07085494
Title: A Double-Blind, Sham-Controlled Trial Investigating Individualized Alpha Neurofeedback Plus Cognitive Training in Paediatric Brain Tumour Survivors
Brief Title: Neurofeedback and Cognitive Training for PBTS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie Wan Yee Tso (Dr), Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HKU_PBTS_NF_CT
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumor, Primary
MeSH Terms: conditions — Brain Neoplasms | interventions — Neurofeedback; Cognitive Training

STUDY DESIGN:
Intervention Model Description: Once eligible participants are enrolled in this study, they will be randomly allocated either to the neurofeedback intervention group or the sham feedback group. Participants in both groups will receive treatment/sham neurofeedback treatment at the same period. Partcipants in both groups receive cognitive training
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A deterministic blinding method will be used. Each participant receives a unique de-identified ID (for example, "NFB001"), which will be processed with a custom hashing function that produces a binary value (0 or 1) with equal probability. This determines whether they receive individualized alpha feedback or sham feedback (by customised algorithm). Throughout the study, only the participant's de-identified ID is visible to researchers, site staff, and participants, thus preserving blinding.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback + Cognitive trianing (Experimental): Participants will receive neurofeedback and cognitive training
  Interventions: Behavioral: neurofeedback; Behavioral: Cognitive Training
- Sham neruofeedback + cognitve trianing (Sham Comparator): Participants will receive sham neruofeedback and cognitive training
  Interventions: Behavioral: Cognitive Training; Behavioral: Sham feedback

INTERVENTIONS:
Behavioral: neurofeedback — - Neurofeedback Training : Feedback is based on individualized alpha band power. Participants see a game-like display (for instance, a plane) that reflects their alpha activity. Excessive EMG (muscle tension) causes performance drops, encouraging relaxation.
  Arms: Neurofeedback + Cognitive trianing
Behavioral: Cognitive Training — - Cogmed Training : Participants complete adaptive tasks focusing on working memory. The difficulty adjusts in real time based on performance.
Behavioral: Sham feedback — The sham neurofeedback protocol was identical to the verum neurofeedback protocol except that the animation (horizontal plane movement) was based on the EEG results of another participant. EMG-based feedback will still be provided for the sham condition
  Arms: Sham neruofeedback + cognitve trianing

SUMMARY:
Brief Summary of the Study:

This study is a prospective, randomized, sham-controlled, triple-blind trial investigating whether combining individualized alpha neurofeedback (NF) with cognitive training (Cogmed) can improve cognitive functioning in pediatric brain tumor survivors (PBTS), a group at risk for persistent cognitive difficulties after cancer treatment. Participants (ages 6-18) who have completed primary cancer therapy and report cognitive problems are randomly assigned to either (1) individualized alpha NF plus Cogmed or (2) sham NF plus Cogmed. Both interventions include eight one-hour sessions over four weeks, with neurofeedback (real or sham) followed by Cogmed training.

The primary outcome is cognitive performance measured by CNS Vital Signs at baseline, post-intervention, and 12-month follow-up. Secondary outcomes include attention, executive function, behavior, and quality of life (measured by SWAN, BRIEF, SDQ, and PedsQL). The study uses rigorous double-blinding and intention-to-treat analysis, with sample size planned at 40-60 participants. Results will determine if individualized alpha NF, when combined with cognitive training, yields greater cognitive and behavioral benefits than cognitive training alone in PBTS.

DETAILED DESCRIPTION:
This study is a prospective, randomized, sham-controlled, double-blind trial designed to evaluate whether individualized alpha neurofeedback (NF) combined with cognitive training (Cogmed) can improve cognitive functioning in pediatric brain tumor survivors (PBTS), who frequently suffer from attention, memory, and executive function difficulties following cancer treatment.

Participants:

The study plans to enroll 40-60 PBTS, aged 6 to 18, who have completed primary cancer treatment at least six months prior and report cognitive difficulties. Major exclusion criteria include severe neurological or psychiatric conditions, interfering medications, and significant sensory or motor deficits.

Design and Intervention:

Participants are randomly assigned (1:1) to one of two groups:

1. Individualized Alpha Neurofeedback + Cogmed (NF Group)
2. Sham Neurofeedback + Cogmed (Sham Group) Both groups participate in eight one-hour sessions over four weeks. Each session includes 30 minutes of neurofeedback (either real, based on each participant's individualized alpha EEG band, or sham, based on pre-recorded EEG data but with identical procedures) followed by 30 minutes of Cogmed cognitive training (adaptive, computerized working memory tasks).

Blinding:

The study is double-blind: both participants and outcome assessors are blinded to group allocation. The neurofeedback software automatically delivers either real or sham feedback according to assignment, maintaining blinding for all involved.

Objectives and Outcome Measures:

The primary objective is to determine whether the combined individualized alpha NF and Cogmed intervention leads to superior improvements in cognitive functioning, measured by CNS Vital Signs, compared to sham NF plus Cogmed. Assessments occur at baseline, immediately post-intervention, and at 12-month follow-up.

Secondary objectives include evaluating changes in attention, executive function, behavior, and quality of life, using validated tools such as the SWAN, BRIEF, SDQ, and PedsQL. The study will also examine neurophysiological changes (qEEG markers) and their relationship to cognitive and behavioral outcomes.

Data Analysis:

Primary and secondary outcomes will be analyzed using mixed linear models to assess group-by-time interactions. An intention-to-treat approach will include all randomized participants, with appropriate methods for handling missing data.

Significance:

This study will clarify whether adding individualized alpha neurofeedback to cognitive training offers additional cognitive and behavioral benefits for pediatric brain tumor survivors, compared to cognitive training alone, using a rigorous double-blind, sham-controlled methodology with a planned sample size of 40-60 participants.

ELIGIBILITY:
Inclusion Criteria:

* - Paediatric brain tumour survivors aged 6 to 18 years
* Completion of primary cancer treatment (for example, surgery, chemotherapy, or radiotherapy) at least six months prior
* Documented or reported cognitive difficulties in attention or executive functioning
* Ability and willingness to attend scheduled sessions over four weeks

Exclusion Criteria:

* - Severe neurological or psychiatric conditions (for example, uncontrolled seizures) that preclude EEG monitoring or completing computer-based training
* Medication regimens that significantly interfere with EEG signals and cannot be safely adjusted
* Severe sensory or motor deficits that would make training infeasible
* Inability or unwillingness to follow study protocol

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
cognitive performance | prior to the intervention, immediate after the interventions & 6 months after the intervention
  cognitive performance as measured by a neurocogntive test battery, CNS VS. the neurocognition Index (NCI) as a compostie score of various cognitive performance will be used

SECONDARY OUTCOMES:
PedsQL (Pediatric Quality of Life Inventory) | prior to the intervention, immediate after the intervention & 6 months after the intervention
  The Pediatric Quality of Life Inventory (PedsQL) is a reliable and validated instrument for assessing health-related quality of life in children and adolescents aged 2-18 years. It consists of 23 items, covering four domains: physical functioning, emotional functioning, social functioning, and school functioning. The PedsQL is designed to measure the impact of various health conditions on children's daily lives and well-being.
SDQ (Strengths and Difficulties Questionnaire) | prior to the intervention, immediate after the intervention 6 months after the intervention
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioral screening questionnaire for children and adolescents aged 2-17 years. It consists of 25 items, covering five domains: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. The SDQ is designed to help identify mental health problems and promote emotional well-being in children and adolescents.
Strengths and Weaknesses of Attention-Deficit/Hyperactivity Symptoms and Normal Behavior Scale (SWAN) | prior to the intervention, immediate after the interventions & 6 months after the intervention
  The Chinese SWAN is a validated instrument for the assessment of ADHD symptoms in Chinese children in Hong Kong. The SWAN questionnaire was originally devised by Swanson et al in 2005 based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for ADHD.
Behaviour Rating Inventory of Executive Function (BRIEF) | prior to the intervention, immediate after the intervention & 6 months after the intervention
  A parent/self-report questionnaire evaluating various components of executive functioning in daily life (for example, planning, working memory, and inhibitory control)

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No